CLINICAL TRIAL: NCT01082315
Title: A Korean Post-Marketing Surveillance Study On Erbitux® (Cetuximab) in Patients With EGFR-expressing, KRAS Wild-type Metastatic Colorectal Cancer
Brief Title: A Korean Post-marketing Surveillance Study on Erbitux® in Patients With Metastatic Colorectal Cancer Refractory to Irinotecan-containing Treatment
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 62202-509 (EMR 62202-551)
Record Dates: First submitted 2010-03-03; First posted 2010-03-08 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal cancer; Neoplasm metastasis; Cetuximab; Erbitux; EGFR
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Erbitux (Cetuximab) — In subjects with mCRC, cetuximab will be used in combination with chemotherapy or as a single agent according to the approved national label as in routine clinical practice. Cetuximab 2mg/ml will be administered intravenously via in-line filtration with an infusion pump, gravity drip or a syringe pump. For the initial dose, the recommended infusion period is 120 minutes and for the subsequent weekly doses, the recommended infusion period is 60 minutes.
  Other Names: Erbitux

SUMMARY:
After consultation with the Korean Health Authorities, the two Post-Authorization Safety Studies EMR 62202-509 (NCT01082315) and EMR 62241-508 (NCT01075828) were combined within one study protocol EMR 062202-551. This Post-Marketing Surveillance Study (PMS) EMR 062202-551 is requested by the Korean Health Authorities to continue monitoring of Erbitux and provide further information about safety and toxicity in clinical practice in at least 900 patients during 6 years.

All data points from the EMR 62202-509 (NCT01082315) and EMR 62241-508 (NCT01075828) remain unchanged in protocol EMR 062202-551. Therefore, the Sponsor has decided not to separately disclose the EMR 062202-551 study titled "A Korean Post-Marketing Surveillance Study On Erbitux® (Cetuximab) in Patients With Locally Advanced or Recurrent and/or Metastatic Squamous Cell Cancer of the Head and Neck (originally EMR 62241-508) and in Patients With EGFR-expressing, KRAS wild-type Metastatic Colorectal Cancer (originally EMR 62202-509)" on clinicaltrials.gov.

DETAILED DESCRIPTION:
This is a post marketing surveillance (PMS), prospective study to collect safety information from more than 600 subjects with epidermal growth factor receptor (EGFR)-expressing, V-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (KRAS) wild-type metastatic colorectal cancer (mCRC) treated with Erbitux as final evaluable cases. This PMS is requested by the Korean Regulatory Authorities because after removal of an orphan drug in Korea, there is a requirement to investigate more than 600 patients during six years, to continue monitoring and provide further information about safety and toxicity in clinical practice.

This PMS study is planned to be conducted within 6 years from the removal date of orphan drug in approximately 50 institutions in Korea.

OBJECTIVES

The objective of the study is to analyse the safety and efficacy information on the use of Erbitux in the market and factors affecting its safety and efficacy.

Primary objective:

* To obtain safety information on the use of Erbitux in subjects with mCRC in terms of frequency and severity of adverse events (AEs)

Secondary objective:

* To gather clinical efficacy information of the treatment

During the PMS period, each subject's background, medical history (surgery, radiotherapy), Erbitux treatment status, concurrent medication, response evaluation, status and reason of discontinuation, all AEs (regardless of the causal relationship to Erbitux), and abnormal results of laboratory tests will be collected from the start of treatment with Erbitux until progressive disease, Erbitux-related intolerable toxicities, death, or withdrawal of Erbitux treatment (whichever occurs first). The primary endpoint, the safety evaluation will be based on all cases treated with Erbitux having received at least one dose. However, for efficacy evaluation, 12 weeks of treatment have to be applied to each subject.

Erbitux will be prescribed to mCRC subjects according to the approved national label as in routine clinical practice, under the supervision of an investigator experienced in the use of antineoplastic medicinal products. Prior to the first infusion, subjects will receive pre-medication with an antihistamine and a corticosteroid. The initial dose of Erbitux is 400 mg/m2 body surface area and the subsequent weekly doses are 250 mg/m2 each administered intravenously via in-line filtration with an infusion pump, gravity drip, or a syringe pump. The recommended infusion period for the initial dose is 120 minutes and for the subsequent weekly doses is 60 minutes with the maximum infusion rate not exceeding 10 mg/min, equivalent to 5 ml/min of Erbitux 2 mg/ml.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are eligible for Erbitux treatment according to the indication in the national label of Erbitux ( i.e. in EGFR expressing, KRAS wild-type mCRC subjects in combination with chemotherapy, or as a single agent in subjects who failed oxaliplatin and irinotecan based therapy and who are intolerant to irinotecan)

Exclusion Criteria:

* Subjects who are not eligible for Erbitux treatment according to the indication in the national label of Erbitux

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with EGFR-expressing, KRAS wild-type mCRC undergoing treatment with Erbitux in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2009-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety | Initial treatment period to final treatment period
  Incidence and severity of all adverse events, regardless of the causal relationship to Erbitux

SECONDARY OUTCOMES:
Clinical efficacy | The evaluation date to show best tumour response during the treatment of Erbitux
  Best tumour response, time to progression of tumour and duration of response with Erbitux treatment; liver metastasis resectability.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea